CLINICAL TRIAL: NCT05493527
Title: Noninvasive High Frequency Oscillatory Ventilation as a Post-extubation Respiratory Support in Preterm Neonates: A Randomized Controlled Trial
Brief Title: Noninvasive High Frequency Oscillatory Ventilation as a Post-extubation Respiratory Support in Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sondos Ahmed Salaheldin Ahmed, Assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD 90/2020
Record Dates: First submitted 2022-08-03; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Infant, Premature, Diseases; Infant, Newborn, Disease; Respiratory Tract Diseases; RDS
Keywords: noninvasive high frequency ventilation; noninvasive ventilation; RDS; post-extubation; preterm; respiratory distress syndrome; noninvasive positive pressure ventilation
MeSH Terms: conditions — Infant, Premature, Diseases; Disease; Respiratory Tract Diseases; Premature Birth; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- noninvasive high frequency oscillatory ventilation (NHFOV) (Experimental): After documenting parental consent, the ventilated infants eligible for extubation were randomly assigned to NHFOV as post extubation noninvasive respiratory support
  Interventions: Device: noninvasive high frequency oscillatory ventilation
- noninvasive positive pressure ventilation (NIPPV) (Active Comparator): After documenting parental consent, the ventilated infants eligible for extubation were randomly assigned to NIPPV as post extubation noninvasive respiratory support
  Interventions: Device: noninvasive positive pressure ventilation

INTERVENTIONS:
Device: noninvasive high frequency oscillatory ventilation — A time-cycled, pressure-limited, and continuous-flow neonatal ventilator (SLE6000; SLE) was used for neonates assigned to the NHFOV group. The settings were as follows:
  1. a frequency of 10 Hertz ( range, 8-12 Hz);
  2. an inspiratory time of 50% (1:1)
  3. an oscillation amplitude of 35 centimeter of water column (cmH2O) (subsequent regulation range, 20-40 cmH2O) Oscillation amplitude would be regulated according to the level of carbon dioxide(CO2). Visible chest oscillation was not necessary because elimination of CO2 during NHFOV could also occur in the upper respiratory airway dead space
  4. Mean airway pressure (MAP) of 10 cm H2O ( range, 7-15) MAP was regulated according to an open lung recruitment strategy
  5. fraction of inspired oxygen (FIO2) regulated from 0.21 to 0.40 in order to maintain saturation from 90% to 95% as determined with a pulse oximeter.
  Arms: noninvasive high frequency oscillatory ventilation (NHFOV)
Device: noninvasive positive pressure ventilation — NIPPV will be delivered by ventilator generating the targeted pressures. Infants will be on:
  1. Peep ranging from 5 to 10 cmH2O,
  2. Peak inspiratory pressure range 15-25 cmH2O
  3. Rate range 40-50 breath/minute
  4. FIO2 regulated from 0.21 to 0.40 in order to maintain saturation from 90% to 95% as determined with a pulse oximeter.
  Arms: noninvasive positive pressure ventilation (NIPPV)

SUMMARY:
A randomized controlled trial comparing Noninvasive high frequency oscillatory ventilation (NHFOV) and Noninvasive positive pressure ventilation (NIPPV) as post-extubation respiratory support in preterm neonates with respiratory distress syndrome(RDS)

DETAILED DESCRIPTION:
The use of noninvasive respiratory support (NRS) has increased in recent decades in Neonatal Intensive Care Unit (NICU) as a means to reduce ventilator-induced lung injury. Various modes of NRS are available and in common use. However despite extensive research, the optimal modality of noninvasive modes remain unknown.

Noninvasive high-frequency oscillatory ventilation (NHFOV) is a relatively new mode. It consists of the application of a continuous distending positive pressure with superimposed oscillations. It is a method of augmenting Continuous positive airway pressure (CPAP) support potentially combining the advantages of both high-frequency oscillatory ventilation and CPAP.

The new NHFOV technique offers improved carbon dioxide (CO2) removal and increased functional residual capacity. The superimposed oscillations of NHFOV are thought to help avoid gas trapping and upregulate mean airway pressure.

This technique is also characterized by lower tidal volume resulting in fewer barotraumas /volutraumas and not needing synchronization. NHFOV was considered a strengthened version of CPAP.

The hypothesis is that NHFOV might be superior to NIPPV as a post-extubation respiratory support strategy to avoid reintubation and subsequent complications and/or sequelae in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm neonates with gestational age ≤ 35 weeks.
2. Neonates that were on invasive mechanical ventilation for at least 48 hours eligible for extubation

Exclusion Criteria:

1. Patients with major upper or lower airway anomalies.
2. Patients with significant congenital anomalies including cardiac, abdominal or respiratory.

Ages: 1 Minute to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Re-intubation rate | 72 hours
  Percentage of Patients who failed weaning on the assigned noninvasive mode and needed reintubation to the total number of patients assigned to that mode.

SECONDARY OUTCOMES:
Days on the assigned non-invasive respiratory support | 8 weeks or till patient discharge which comes first
  To document number of days on the assigned non-invasive respiratory support
Days on supplemental oxygen | 8 weeks or till patient discharge which comes first
  To document number of days on supplemental oxygen
Duration of admission | 8 weeks or till patient discharge which comes first
  To document total number of days of admission
Mortality rate | 8 weeks or till patient death which comes first
  To document incidence of mortality during hospitalization
Lung ultrasound score | Before extubation and after 2 hours on assigned mode
  lung ultrasound was performed to all patients before extubation and 2 hours after extubation to assess lung aeration. Score ranges from 0 to 18 .Higher score indicates worse lung aeration.
Co2 change | Before extubation and after 2 hours on assigned mode
  Co2 change in patients on assigned mode using venous blood gases performed before extubation and 2 hours after.
Oxygen requirement | Before extubation and after 2 hours on assigned mode
  Fraction of inspired oxygen required to patients on assigned mode
Incidence of feeding intolerance | 8 weeks or till patient weaning from assigned mode which comes first
  Percentage of Patients who developed feeding intolerance on the assigned noninvasive mode to the total number of patients assigned to that mode.
Days to reach full intake | 8 weeks or till patient discharge which comes first
  Number of days needed by each patient to reach full intake
Intracranial hemorrhage | 8 weeks or till patient weaning from assigned mode which comes first
  Percentage of patients developing intracranial hemorrhage on the assigned noninvasive mode to the total number of patients assigned to that mode.
Pneumothorax | 8 weeks or till patient weaning from assigned mode which comes first
  Percentage of patients developing pneumothorax on the assigned noninvasive mode to the total number of patients assigned to that mode.
Incidence of occurrence of Nasal trauma | 8 weeks or till patient weaning from assigned mode which comes first
  Percentage of patients developing nasal trauma on the assigned noninvasive mode to the total number of patients assigned to that mode.
incidence of bronchopulmonary dysplasia | 8 weeks or till patient discharge which comes first
  Need for supplemental oxygen for at least 28 days, percentage of these patients on the assigned noninvasive mode to the total number of patients assigned to that mode.
Severity of respiratory distress | Before extubation and and after 2 hours on assigned mode
  Assessment of work of breathing on assigned mode by Downe 's score. Score ranges from 0 till 10 . Higher score indicates worse work of breathing.
Need for Postnatal Steroids | 8 weeks or till patient discharge which comes first
  Percentage of patients who needed postnatal steroids administration
Chest x ray change | Before extubation and and after 2 hours on assigned mode
  Chest x ray grading of RDS performed to patient before and after the assigned mode to compare lung aeration degree.

CONTACTS AND LOCATIONS:
Locations (1):
- Neonatal Intensive Care Units (NICUs), Ain Shams University, Cairo, Abbasia, Egypt